CLINICAL TRIAL: NCT00343161
Title: A Randomized, Open, Parallel-group, Multi-national, Multi-centre, Phase IV Study to Evaluate the Efficacy of Three Different Patient Management Strategies With and Without Esomeprazole 20 mg During a 3 Months Maintenance Phase Following an Initial 4-weeks Acute Treatment Phase in Subjects With Symptoms Thought to be GERD Related
Brief Title: Symptom Adapted Therapy in GERD Patients
Acronym: SYMPATHY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00109; SYMPATHY; EudraCT-No. 2006-001316-76
Record Dates: First submitted 2006-06-20; First posted 2006-06-22 (Estimated); Last update posted 2011-01-24 (Estimated); Status verified 2011-01

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: Nexium
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

INTERVENTIONS:
Drug: esomeprazole
Drug: Gelusil-Lac (Aluminum hydroxide gel,magnesium trisilicate)

SUMMARY:
The purpose of the study is to determine whether a maintenance treatment over 12 weeks with esomeprazole 20 mg daily will sufficiently give control over GERD symptoms and how it compares either with an on-demand therapy with esomeprazole 20 mg or an as needed therapy (wait and see regimen) with rescue medication only (antacid), following a 4-weeks acute treatment phase with either esomeprazole 20 mg or esomeprazole 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Patients who seek medical advice in primary care for symptoms thought to be GERD-related

Exclusion Criteria:

* Clinical GERD diagnosis/treatment within last 3 month
* History of severe esophagitis (i.e. LA grade C or D)
* Previous anti-reflux surgery
* History of drug abuse
* Female patients who are pregnant or lactating or at risk of pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 441
Dates: Start 2006-08; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of three different long-term treatment strategies in primary care setting
To compare treatments separately within different levels of symptom load according to clinical judgement at baseline
Number of 'treatment failures' used as primary outcome variable.

SECONDARY OUTCOMES:
To evaluate whether the Reflux Disease Questionnaire (RDQ)used in primary care setting adds value to clinical judgement in assessing baseline symptom load
Evaluate whether the RDQ facilitates the decision on appropriate acute and maintenance treatment strategy
To assess the additional impact of a concomitant low dose acetylsalicylic acid (ASA) therapy during acute and maintenance phase with regard to efficacy
To evaluate whether there is a difference between treatment strategies with regard to patient satisfaction during maintenance phase using the GERD Impact Scale

CONTACTS AND LOCATIONS:
Overall Officials: Michael Höcker, MD, Study Director — AstraZeneca Germany; Joachim Labenz, MD, Principal Investigator — Evan. Jung-Stilling-Krankenhaus, Siegen, Germany
Locations (96):
- Germany (96):
  - Research Site, Aiterhofen
  - Research Site, Ansbach
  - Research Site, Apolda
  - Research Site, Bad Bramstedt
  - Research Site, Bad Frankenhausen
  - Research Site, Bad Salzuflen
  - Research Site, Bad Schwartau
  - Research Site, Baden-Baden
  - Research Site, Bergkamen
  - Research Site, Bergrheinfeld
  - Research Site, Berlin
  - Research Site, Bielefeld
  - Research Site, Bietigheim-Bissingen
  - Research Site, Blankenhain
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Burgwedel
  - Research Site, Cologne
  - Research Site, Dahn
  - Research Site, Deggendorf
  - Research Site, Deggingen
  - Research Site, Dresden
  - Research Site, Duisburg
  - Research Site, Düsseldorf
  - Research Site, Engstingen
  - Research Site, Erfurt
  - Research Site, Erlangen
  - Research Site, Essen
  - Research Site, Ettlingen
  - Research Site, Falkensee
  - Research Site, Freudenberg
  - Research Site, Fürstenwalde
  - Research Site, Garching
  - Research Site, Gärtringen
  - Research Site, Gefell
  - Research Site, Gera
  - Research Site, Gladbeck
  - Research Site, Goch
  - Research Site, Görlitz
  - Research Site, Greven
  - Research Site, Hamm
  - Research Site, Hammelburg
  - Research Site, Heidelberg
  - Research Site, Heilbronn
  - Research Site, Heiligenstadt
  - Research Site, Heroldsberg
  - Research Site, Herrischried
  - Research Site, Hoyerswerda
  - Research Site, Ilmenau
  - Research Site, Isernhagen-Süd
  - Research Site, Kehl
  - Research Site, Kirchlengern
  - Research Site, Krefeld
  - Research Site, Kronach
  - Research Site, Landau
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, Lohfelden
  - Research Site, Löbau
  - Research Site, Löhne
  - Research Site, Lübbecke
  - Research Site, Lübeck
  - Research Site, Magstadt
  - Research Site, Mülsen
  - Research Site, Münster
  - Research Site, Netphen
  - Research Site, Neuss
  - Research Site, Oberwiesenthal
  - Research Site, Oettingen in Bayern
  - Research Site, Otterbach
  - Research Site, Pforzheim
  - Research Site, Plettenberg
  - Research Site, Porta Westfalica
  - Research Site, Rehmsdorf
  - Research Site, Reinfeld
  - Research Site, Rheinmünster-Greffern
  - Research Site, Saarbrücken
  - Research Site, Schnaittenbach
  - Research Site, Schwerte
  - Research Site, Siegen
  - Research Site, Spalt
  - Research Site, Stutensee
  - Research Site, Sulzheim
  - Research Site, Teterow
  - Research Site, Thurnau
  - Research Site, Uhingen
  - Reseach Site, Urspringen
  - Research Site, Viersen
  - Research Site, Vilshofen
  - Research Site, Waghäusel
  - Research Site, Walsrode
  - Research Site, Weinheim
  - Research Site, Weißwasser
  - Research Site, Wesseling
  - Research Site, Wuppertal
  - Research Site, Zwickau